CLINICAL TRIAL: NCT01000532
Title: Pilot Study to Compare Steroid (SIELLO T/JT) Versus Non-Steroid Pacing Leads (BPPU T/JT)
Brief Title: SIELLO Pilot Study for Comparison of Steroid Versus Non-Steroid Pacing Leads
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 47-1
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Arrhythmias, Cardiac
Keywords: steroid, leads, threshold, pacemaker
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pacemaker therapy
  Interventions: Device: SIELLO JT/T; Device: Pacemaker therapy; Device: BPPU JT/T

INTERVENTIONS:
Device: SIELLO JT/T — Implantation of SIELLO and BPPU pacemaker leads
  Other Names: BPPU JT/T
Device: Pacemaker therapy — Pacemaker therapy
Device: BPPU JT/T — Implantation of SIELLO and BPPU pacemaker leads

SUMMARY:
This investigation is designed to demonstrate the clinical efficacy and safety of the low-dose drug of the SIELLO leads in comparison to the non-steroid BPPU leads in a clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for pacemaker therapy
* Understand the nature of the procedure
* Give informed consent
* Able to complete all testing required by the clinical protocol
* Available for follow-up visits on a regular basis at the investigational site

Exclusion Criteria:

* Meet none of the pacemaker indications
* Meet one or more of the contraindications
* Have a life expectancy of less than six months
* Cardiac surgery in the next six months
* Enrolled in another cardiac clinical investigation
* Have other medical devices that may interact with the implanted pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard pacemaker indication who are refered to the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Béla Merkely, Professor, Principal Investigator — Semmelweis University Heart Center, Budapest, Hungary
Locations (1):
- Semmelweis University, Budapest, Hungary

REFERENCES:
- [Derived] Kutyifa V, Zima E, Molnar L, Kuehne C, Theiss S, Herrmann G, Geller L, Merkely B. Direct comparison of steroid and non-steroid eluting small surface pacing leads: randomized, multicenter clinical trial. Cardiol J. 2013;20(4):431-8. doi: 10.5603/CJ.2013.0103. PMID 23913463